CLINICAL TRIAL: NCT00204425
Title: Effect of Combined Exercise Therapy and Isoflavone Supplementation on Prevention of Osteoporosis
Brief Title: Effect of Exercise Training and Soy-based Nutritional Supplementation on Prevention of Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Factorial | Masking: Quadruple
Other Study IDs: Bio 03-1077; 124322 FRN68095
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2011-09

CONDITIONS: Osteoporosis; Osteopenia
Keywords: Osteoporosis; Bone; Exercise; Soy; Isoflavone; Phytoestrogen; Menopause; Lipids
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): exercise/soy isoflavone
  Interventions: Dietary Supplement: exercise/soy isoflavone
- 2 (Experimental): exercise/isoflavone placebo
  Interventions: Dietary Supplement: exercise/soy isoflavone
- 3 (Experimental): exercise placebo/soy isoflavone
  Interventions: Dietary Supplement: exercise/soy isoflavone
- 4 (Placebo Comparator): exercise placebo/isoflavone placebo
  Interventions: Dietary Supplement: exercise/soy isoflavone

INTERVENTIONS:
Dietary Supplement: exercise/soy isoflavone — Exercise 6 days per week, 90 mg/day aglycone isoflavone Exercise placebo (stretching), isoflavone placebo
  Other Names: Archer Daniels Midland

SUMMARY:
The purpose of the study is to determine the effectiveness of combining exercise training (i.e. weight lifting and walking) and dietary supplementation with a soy-based nutritional supplement for increasing bone mineral density. We hypothesize that the exercise training and soy-based supplement will be additive for increasing bone mineral density.

DETAILED DESCRIPTION:
Exercise training is effective for increasing bone mineral density and preventing osteoporosis, but the effects are small. When estrogen replacement is given to post-menopausal women the effectiveness of exercise training for improving bone mineral density is increased. Currently many women are concerned about the risks of taking hormone-replacement therapy and are seeking alternative therapies. The purpose of our study therefore is to use an estrogen-like dietary supplement derived from soy called a phytoestrogen (soy isoflavone) combined with exercise training for improving bone mineral density.

Comparisons: Four groups are being compared: 1) Exercise training (i.e. weight lifting 2 times per week and walking 4 times per week) plus soy isoflavone (90 mg aglycone equivalents per day); 2) Exercise training plus placebo; 3) Exercise placebo (flexibility exercises four times per week) plus soy isoflavone; 4) Exercise placebo plus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal women

Exclusion Criteria:

* Diagnosed osteoporotic
* Previous fragility fractures
* Previous breast cancer
* Previous endometrial cancer
* Taken bisphosphonates in past 12 months
* Taken hormone replacement therapy in past 12 months
* Taken selective estrogen receptor modulators in past 12 months
* Taken parathyroid hormone in past 12 months
* Taken calcitonin in past 12 months
* Currently taking corticosteroids
* Currently taking a thiazide diuretic
* Crohn's Disease
* Cushing Disease
* Allergy to soy
* Severe osteoarthritis
* Currently participating in vigorous exercise

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2004-12; Primary Completion 2007-12 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Lumbar spine bone mineral density at 12 and 24 months | 2 years

SECONDARY OUTCOMES:
Bone mineral density of the proximal femur at 12 and 24 months. | 2 years
Bone mineral density of the whole body at 12 and 24 months. | 2 years
Bone quality of the radius and tibia (ultrasound) at 12 and 24 months. | 2 years
Geometry of the proximal femur at at 12 and 24 months. | 2 years
Lean tissue mass at 12 and 24 months. | 2 years
Fat mass at 12 and 24 months. | 2 years
Body mass index at 12 and 24 months. | 2 years
Waist girth at 12 and 24 months. | 2 years
Blood lipids at 12 and 24 months. | 2 years
Muscular strength at 12 and 24 months. | 2 years
Self-paced walking ability at 12 and 24 months. | 2 years
Balance at 12 and 24 months. | 2 years
Flexibility at 12 and 24 months. | 2 years
Breast density at 24 months | 2 years
Endometrial thickness at 24 months. | 2 years
Menopausal symptoms at 3, 6, 9, 12, 15, 18, 21, and 24 months. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Philip D Chilibeck, PhD, Principal Investigator — University of Saskatchewan; H J Biem, M.D., Study Director — University of Saskatchewan; Allison Case, M.D., Study Director — University of Saskatchewan; Olufemi Olantunbosun, M.D., Study Director — University of Saskatchewan; Roger Pierson, PhD, Study Director — University of Saskatchewan; Susan Whiting, PhD, Study Director — University of Saskatchewan; Punam Pahwa, PhD, Study Director — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Background] Chilibeck PD. Exercise and estrogen or estrogen alternatives (phytoestrogens, bisphosphonates)for preservation of bone mineral in postmenopausal women. Can J Appl Physiol. 2004 Feb;29(1):59-75. doi: 10.1139/h04-006. PMID 15001805